CLINICAL TRIAL: NCT00460291
Title: Pilot Study to Asses the Function and Patency of Polyester-Coated Composite Bypasses From Autologous Varicose Veins
Acronym: PROVENA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ProVena
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2007-10-03 (Estimated); Status verified 2007-10

CONDITIONS: Peripheral Arterial Disease; Peripheral Bypass Surgery; Bypass From Autologous Varicose Vein; External Graft Support
Keywords: PAD; vein bypass; supported varicose veins
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Implantation of the ProVena vein graft during bypass surgery

SUMMARY:
If patients need to undergo bypass surgery, either an autologous vein can be used as bypass or, if there are no suitable veins are available, a prosthetic graft can be implanted. Varicose veins normally are judged not to be suitable as bypass. The ProVena vein support, made from polyester, is considered to strengthen varicose veins so that they they become suitable as bypass. Thereby, the advantages of an autologous bypass and the stability of polyester material can be combined.

Patients that take part in the trial recieve an autologus bypass with a varicose vein, coated with ProVena. They are followed up at 3 and 6 months after implantation of a ProVena-coated bypass via duplex-sonography to assess the graft patency.

DETAILED DESCRIPTION:
The ProVena trial is a non-randomised multi-centre trial, aiming to assess the suitability of the ProVena vein support.

Currently, autologous veins are preferred to prosthetic grafts (Klinkert et al. 2004), but they are not considered to be suitable if they are varicose.

Some early data indicate that these veins can be used if an external support is applied (Moritz et al. 1993, 1992, Neufang et al. 2003). The proVena vein graft has been tested in animal experiments. All bypasses showed a reduced intima hyperplasia, no disadvantages were found. Nevertheless, as a ProVena-coated bypass cannot be regarded as completely autologus, it is necessary whether the coating does not increase the risk of

* infections
* scar formation, reducing the patency
* higher incidence of seroma

ProVena is made from polyester filaments, similar to the material used for prosthetic grafts. As the material is used since years in peripheral bypass surgery, we do not expect increased risks.

It is planned to include 50 Patients in 10 centres. Patients can be included if they match the eligibility criteria, need to undergo peripheral bypass surgery and have varicose veins normally not suitable to form a bypass graft. If patients agree to take part and give informed consent, baseline data are collected and the surgery is protocolled. Patients are followed up after 3 ands six months by duplex sonography. The inflammation parameters are detected via analysis of a blood sample. Main endpoints and secondary endpoints are as follows:

Main endpoints:

* Infection rate
* primary patency
* primary assisted patency
* secondary patency

Secondary endpoints:

* complication rate
* occurence of bypass stenosis
* time needed for preparation of the bypass vein
* technical success i. e. successful implatation of the ProVena Graft

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 years 18 Jahre.
* informed consent has been given and patients is complient to protocol
* patient needs femoro-distal bypass surgery
* only varicose ektatic veins are available
* Bypass diameter > 5mm proximal and > 4mm distal.

Exclusion Criteria:

* aged < 18 years
* patient unable to take part in the follow-up
* known sensibility to polyester
* patient not expected to survive the next 12 months due to significant comorbidities
* HIV-infection
* Patient suffering from a floriding infection at the time of inclusion
* infection or colonisation with MRSA
* pregnancy
* use of immunosuppresive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-06; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
infection rate
primary patency
primary assisted patency
secondary patency

SECONDARY OUTCOMES:
occurrence of complications
occurence of stenoses
time needed for preparation of the bypass vein
technical success

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schmitz-Rixen, MD, Professor, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (11):
- Germany (11):
  - Charité, Berlin
  - Cologne University Hospital, Cologne
  - Kath. Kliniken Essen-Nord, Essen
  - Nordwestkrankenhaus Frankfurt, Frankfurt
  - Frankfurt University Hospital, Frankfurt am Main
  - Municipal Hospital Karlsruhe, Karlsruhe
  - Frankenwaldklinik Kronach gGmbH, Kronach
  - Mainz University Hospital, Mainz
  - Municipal Hospital, Mühldorf
  - St. Franziskus Hospital, Münster
  - Verbundkrankenhaus Bernkastel/Wittlich, Wittlich

REFERENCES:
- [Background] Klinkert P, Post PN, Breslau PJ, van Bockel JH. Saphenous vein versus PTFE for above-knee femoropopliteal bypass. A review of the literature. Eur J Vasc Endovasc Surg. 2004 Apr;27(4):357-62. doi: 10.1016/j.ejvs.2003.12.027. PMID 15015183
- [Background] Moritz A, Grabenwoger F, Raderer F, Ptakovsky H, Magometschnigg H, Ullrich R, Staudacher M. Use of varicose veins as arterial bypass grafts. Cardiovasc Surg. 1993 Oct;1(5):508-12. PMID 8076087
- [Background] Moritz A, Grabenwoger F, Raderer F, Ptakovsky H, Staudacher M, Magometschnigg H, Ullrich R, Wolner E. Mesh tube--constricted varicose veins used as bypass grafts for infrainguinal arterial reconstruction. Arch Surg. 1992 Apr;127(4):416-20. doi: 10.1001/archsurg.1992.01420040058010. PMID 1558494
- [Background] Neufang A, Dorweiler B, Espinola-Klein C, Reinstadler J, Kirsch D, Schmiedt W, Oelert H. External reinforcement of varicose veins with PTFE prosthesis in infrainguinal bypass surgery -- clinical results. Thorac Cardiovasc Surg. 2003 Apr;51(2):62-6. doi: 10.1055/s-2003-38985. PMID 12730812